CLINICAL TRIAL: NCT06509061
Title: "I am a Physically Active Person!": A Randomized Controlled Trial Aimed to Increase Levels of Physical Activity Self-Definition and Physical Activity Among a Sample of Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Research Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E2013:120
Record Dates: First submitted 2024-06-28; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity Self-Definition; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants were told that they were in one of two informational sessions; they were not told if they were in the intervention or the control group. Researchers sending the surveys to participants' emails were also blinded to the condition. Intervention facilitators who were presenting the material were necessarily aware of the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASD Intervention (Experimental): 6 week 30-45 minute psychoeducation sessions that delivered content on the variables within the Physical Activity Self-Definition Model. The first session was an introductory session and each one that followed focused on one of the direct or indirect determinants of the model: perceived enjoyment, perceived wanting, perceived commitment, perceived trying, perceived ability (all relating to physical activity). Group activities such as worksheets and discussion were carried out during the session.
  Interventions: Other: Physical Activity Self-Definition
- Attention Control (Active Comparator): 6 week 30-45 minute educational sessions that delivered content on general health behaviour. After the introductory session, each week, one of five general health behaviours were covered: balanced diet, sleep, reducing sedentary behaviour, mental/spiritual health and self-compassion/cultivating positive health behaviours. Group activities such as worksheets and discussion were carried out during the session.
  Interventions: Other: Control

INTERVENTIONS:
Other: Physical Activity Self-Definition — 6 week behavioural change program designed to increase PASD and PA
  Arms: PASD Intervention
Other: Control — 6 week program designed to as an attention control, delivering content on general health behaviour.
  Arms: Attention Control

SUMMARY:
This explanatory sequential mixed methods study investigated if an intervention can increase the physical activity identity and physical activity (PA) of inactive individuals. The intervention condition focused on increasing participant's physical activity self-definition (PASD) through educational sessions and group discussions on the five direct and indirect determinants of PASD (perceived enjoyment, perceived wanting, perceived commitment, perceived trying, perceived ability). The control condition was given general health behaviour education sessions. Researchers conducted interviews with some of the participants after the intervention was completed.

ELIGIBILITY:
Inclusion Criteria:

* Must be insufficiently active (<150 minutes of moderate-vigorous PA per week)
* Scored below the mean in PASD
* Medically safe to participate in PA
* Intention to engage in PA over the next 6 weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Physical Activity Self-Definition | Measured pre-intervention, 5 weeks later at intervention end and 4 weeks post intervention
  Measured with a 4-item questionnaire using a 7-point Likert scale (1= strongly disagree; 7 = strongly agree)
ActiGraph Accelerometers | Measured pre-intervention, 5 weeks later at intervention end and 4 weeks post intervention
  Weekly sedentary, light, moderate, and vigorous physical activity minutes were measured using accelerometers, worn at the hip for 7 day during waking hours.

IPD SHARING:
Plan to Share IPD: No
We do not have ethics approval to share data